CLINICAL TRIAL: NCT06701188
Title: Supportive Training After Cardiac Rehabilitation Including Virtual Engagement: The STRIVE Study
Brief Title: Supportive Training After Cardiac Rehabilitation Including Virtual Engagement
Acronym: STRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Davis (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-41119; 1R01HL171287 (NIH)
Record Dates: First submitted 2024-11-05; First posted 2024-11-22 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Adherence to Physical Activity After Completing Cardiac Rehabilitation (CR) in Older Adults
Keywords: Cardiac rehabilitation; Adherence; Cardiovascular disease; m-Health; Physical Activity; Social support
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile App Alone (No Intervention): Mobile app control group. Exposure time will be similar between participants in both the intervention and control groups as both will have: (1) continuous access to the app for self-monitoring of exercise, blood pressure, and weight; (2) weekly "push" text messages with access to a library of educational content for learning that is self-paced on the app over 6 months; and (3) assigned 1 video per month on a variety of health topics related to older adults via the app that match exposure time (approximately 20-30 minutes) with the intervention group. The videos will be created or resourced from reputable organizations. The coach will send weekly short one-way messages on goals, self-management, etc. that the intervention group will also receive. The 1-way messages will be derived from a bank of 210 secondary prevention messages for CVD (PA, nutrition, stress management, heart disease facts, etc.).
- Mobile app + Social (Experimental): The intervention group will also receive Virtual coaching. The coach will evaluate goals, progress, facilitators (use of the buddy system) and challenges with an emphasis on forming healthy PA habits that will be sustained long-term over the life course. Social support: For the social support component, we will provide ground rules for communication (e.g., positive posts, use of "likes", comments, etc.). Groups will be comprised of 4-6 participants with consecutive recruitment.
  Interventions: Behavioral: Virtual Coaching and social support

INTERVENTIONS:
Behavioral: Virtual Coaching and social support — The investigators propose a randomized clinical trial (RCT) of a virtual coaching and social support intervention that integrates evidence- and theory-based approaches to build self-efficacy, self-regulation, and perceived social support after cardiac rehabilitation (CR) to improve physical activity, psychosocial, social cognitive, and clinical outcomes, delivered via a social networking platform (Trainerize). Our intervention will also include goal setting for exercise and tailored feedback by our qualified intervention team.
  Arms: Mobile app + Social

SUMMARY:
The proposed research seeks to determine whether virtual coaching and social support focusing on key social cognitive factors will be an effective strategy for maintaining physical activity (PA) after completing cardiac rehabilitation (CR). Despite the well-documented benefits of CR, only 15-50% of individuals continue to exercise 6 months after completing CR.4-6 Thus, after 36 sessions (typically 12 weeks), many patients are left without the support necessary to sustain physical activity (PA) and prevent adverse secondary cardiac events. Though previous research has explored interventions to sustain PA after CR, many studies have been lacking in a theoretical basis, objective measurement of PA, measurement, and analysis of psychosocial and social cognitive factors, and long-term impact on clinical outcomes. Low-cost, pragmatic approaches to maintaining PA after CR is urgently needed for older adults, and virtual technologies offer promising solutions to promote adherence to PA. The three specific aims of the project are to: 1) determine the effect of virtual coaching and social support on adherence to PA (measured by objective step counts) in the intervention vs. control groups; secondary measures will be amount of sedentary time, functional fitness, and self-reported exercise; 2) determine the effect of virtual coaching and social support on psychosocial and social cognitive factors in the intervention vs. control groups; 2a) evaluate the extent to which psychosocial and social cognitive factors mediate the effect of the intervention on PA adherence; 3) examine differences in cardiovascular (CVD) risk factors (blood pressure, lipids, HbA1c, BMI) between groups.

DETAILED DESCRIPTION:
The investigators propose a randomized clinical trial in which the "STRIVE" control group will receive the Trainerize mobile app for (1) daily self monitoring of exercise, blood pressure, and weight; (2) education via weekly text messages; and (3) assigned monthly videos on various health topics. The "STRIVE +" intervention group will receive the same app for self-monitoring and education via text messages as the control group PLUS individually-tailored virtual coaching with goal-setting and social support/networking. Our specific aims are to:

Aim 1: Determine the effect of virtual coaching and social support on adherence to physical activity (PA; measured by objective step counts) in the intervention vs. control groups; secondary measures will be amount of sedentary time, functional fitness, and self-reported exercise.

Hypothesis 1: The intervention group will have more PA steps and self-reported exercise, less sedentary time, and higher functional fitness compared to the control group.

Aim 2: Determine the effect of virtual coaching and social support on psychosocial and social cognitive factors in the intervention vs. control groups.

Hypothesis 2: The intervention group will have lower depression/loneliness and higher self-efficacy/perceived social support compared to the control group.

Aim 2a: Evaluate the extent to which psychosocial and social cognitive factors mediate the effect of the intervention on PA adherence. Hypothesis 3: Lower depression/loneliness and higher perceived social support will mediate the effect of the intervention on PA adherence.

Aim 3: Examine differences in CVD risk factors (blood pressure, lipids, HbA1c, BMI) between groups. H: The intervention group will have better control of risk factors at 6, 12, and 18 months compared to control.

ELIGIBILITY:
Study population: We will recruit 286 older adults who are 55 years and older with qualifying diagnoses for cardiac rehabilitation (CR).

Inclusion Criteria:

1. ≥ 55 years of age
2. History of CVD that qualified patient for CR (myocardial infarction, percutaneous coronary intervention, coronary artery bypass grafting, heart failure, valve replacement, etc.)
3. Adherence (>50% of sessions for ≥1 month) to outpatient Phase II CR and pending completion

Exclusion Criteria:

1. Participation in Phase III CR (optional extended CR after outpatient Phase II CR for those who pay out-of-pocket)
2. Cognitive impairment (per Mini-Cog assessment tool with score 0-2)
3. Lack of English or Spanish proficiency/literacy
4. Clinical conditions including:

   1. Unstable arrhythmias, aortic stenosis, thrombophlebitis, dissecting aneurysm or symptomatic anemia
   2. Active infection
   3. Uncontrolled hypertension: resting systolic >180 mmHg, diastolic >100 mmHg
   4. Decompensated heart failure, NYHA Class III-IV
   5. Current unstable angina
   6. 2nd or 3rd degree heart block or exercise induced arrhythmias

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Step counts | At baseline, 3, and 6 months
  The primary outcome of step counts will be collected from the Fitbit. Baseline measurements will be compared to repeated measures over time. Patients will wear the Fitbit for the 1-week run-in period before randomization then will wear it for 2 weeks at the end of month 3 and again at the end of month 6.

SECONDARY OUTCOMES:
Physical Activity, barriers and sedentary time: Rapid Assessment of Physical Activity scale | Baseline, 3, 6, and 12 months
  This 9-item questionnaire assesses self-reported physical activity (higher score indicates higher activity, scored 0-9)
Physical Activity, barriers and sedentary time: Exercise Barriers Scale | Baseline, 3, 6, and 12 months
  This 14-item questionnaire assesses exercise barriers. (Higher score associated with more positive perceptions of exercise, scored 14-56)
Physical Activity, barriers and sedentary time: Self-reported sedentary time | Baseline, 3, 6, and 12 months
  The modified 1-item International Physical Activity Questionnaire assesses self-reported sedentary time (minutes/hours per day)
Functional fitness tests: sit-to-stand | Baseline, 3, 6, and 12 months
  Investigators will assess the functional fitness outcomes by performing the 1 min sit-to-stand test (number of times from sitting to standing and back again within 60 seconds)
Functional fitness tests: 2 minute step test | Baseline, 3, 6, and 12 months
  Investigators will assess the functional fitness outcomes by performing the 2-minute step test (number of times knee raised to designated position within 2 minutes)
Functional fitness tests: dumbbell curl test | Baseline, 3, 6, and 12 months
  We will assess the functional fitness outcomes by performing the dumbbell curl test (number of dumbbell curls within 30 seconds)
Psychosocial factors: Depression | Baseline, 3, 6, and 12 months
  The 8-item Patient Health Questionnaire (PHQ-8) will be used to measure depressive symptoms (higher score associated worse depression, scored 0-24)
Psychosocial factors: Loneliness | Baseline, 3, 6, and 12 months
  Social Isolation Short Form 4a survey (PROMIS) featuring 4 questions adapted from the 20-question UCLA Loneliness Scale (Higher score associated with greater feelings of loneliness/isolation, scored 4-20)
Social cognitive factors: Self-efficacy | Baseline, 3, 6, and 12 months
  The 9-item Self-efficacy for Exercise scale uses components of Social Cognitive Theory (higher score associated higher self-efficacy, scored 0-90)
Social cognitive factors: Self-regulation | Baseline, 3, 6, and 12 months
  The 12-item Physical Activity Self-Regulation scale (PASR-12) has 6 sub-scales including self-monitoring, goal-setting, eliciting social support, reinforcement, time management, and relapse prevention (higher score associated with higher self-regulation, scored 12-60)
Social cognitive factors: Perceived social support | Baseline, 3, 6, and 12 months
  The 12-item Multidimensional Scale of Perceived Social Support includes 3 subscales: family, friends, and significant other (higher score associated with higher perceived social support, scored 12-84)
CV risk factors: hyperlipidemia | Baseline, 3, 6, 12, and 18 months
  Lipids assessed from blood test results from the electronic medical record (EMR)
CV risk factors: hypertension | Baseline, 3, 6, 12, and 18 months
  Hypertension assessed from blood pressure results from the electronic medical record (EMR)
CV risk factors: diabetes | Baseline, 3, 6, 12, and 18 months
  Hemoglobin A1c assessed from blood test results from the electronic medical record (EMR)
CV risk factors: obesity | Baseline, 3, 6, 12, and 18 months
  BMI assessed from the electronic medical record (EMR)

OTHER OUTCOMES:
Cardiac events and rehospitalization trends: Cardiac events | 3, 6, 12, and 18 months
  Number of occurrences of cardiac events (e.g., myocardial infarction, revascularization) collected via EMR/self-report
Cardiac events and rehospitalization trends: Rehospitalizations | 3, 6, 12, and 18 months
  Number rehospitalizations (cardiac and non-cardiac causes) collected via EMR/self-report

CONTACTS AND LOCATIONS:
Overall Officials: Linda Park, PhD, NP, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leon AS, Franklin BA, Costa F, Balady GJ, Berra KA, Stewart KJ, Thompson PD, Williams MA, Lauer MS; American Heart Association; Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention); Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity); American association of Cardiovascular and Pulmonary Rehabilitation. Cardiac rehabilitation and secondary prevention of coronary heart disease: an American Heart Association scientific statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Cardiac Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity), in collaboration with the American association of Cardiovascular and Pulmonary Rehabilitation. Circulation. 2005 Jan 25;111(3):369-76. doi: 10.1161/01.CIR.0000151788.08740.5C. PMID 15668354
- [Background] Ades PA, Maloney A, Savage P, Carhart RL Jr. Determinants of physical functioning in coronary patients: response to cardiac rehabilitation. Arch Intern Med. 1999 Oct 25;159(19):2357-60. doi: 10.1001/archinte.159.19.2357. PMID 10547176
- [Background] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Background] Hellman EA. Use of the stages of change in exercise adherence model among older adults with a cardiac diagnosis. J Cardiopulm Rehabil. 1997 May-Jun;17(3):145-55. doi: 10.1097/00008483-199705000-00001. PMID 9187980
- [Background] Moore SM, Charvat JM, Gordon NH, Pashkow F, Ribisl P, Roberts BL, Rocco M. Effects of a CHANGE intervention to increase exercise maintenance following cardiac events. Ann Behav Med. 2006 Feb;31(1):53-62. doi: 10.1207/s15324796abm3101_9. PMID 16472039
- [Background] Elnaggar A, von Oppenfeld J, Whooley MA, Merek S, Park LG. Applying Mobile Technology to Sustain Physical Activity After Completion of Cardiac Rehabilitation: Acceptability Study. JMIR Hum Factors. 2021 Sep 2;8(3):e25356. doi: 10.2196/25356. PMID 34473064
- [Background] Stafford M, von Wagner C, Perman S, Taylor J, Kuh D, Sheringham J. Social connectedness and engagement in preventive health services: an analysis of data from a prospective cohort study. Lancet Public Health. 2018 Sep;3(9):e438-e446. doi: 10.1016/S2468-2667(18)30141-5. Epub 2018 Aug 22. PMID 30143472
- [Background] Holt-Lunstad J, Robles TF, Sbarra DA. Advancing social connection as a public health priority in the United States. Am Psychol. 2017 Sep;72(6):517-530. doi: 10.1037/amp0000103. PMID 28880099